CLINICAL TRIAL: NCT06093880
Title: Observational, Non-controlled, Prospective Clinical Investigation to Evaluate Long-term Safety and Performance of Mini 4 Ready Intraocular Lenses in Cataract Patients
Brief Title: Observational, Prospective Clinical Investigation on Mini 4 Ready Intraocular Lens
Status: Active, not recruiting | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 054/SI
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cataract
Keywords: Monofocal IOL; Monofocal intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: monofocal intraocular lens — monofocal aspheric hydrophilic-hydrophobic intraocular lens

SUMMARY:
Cataract surgery presents an extremely high success rate in improving vision and quality of life and it is currently the most commonly performed ophthalmic surgery, especially considering its growing utility in the aging population (e.g., more than 20 million worldwide underwent the procedure in 2015); it is possible to affirm that benefits clearly outweigh risks.

However, although cataract surgery is highly effective and relatively safe, owing to the enormous numbers, even uncommon surgical complications could potentially harm the patients. For this reason, it is essential to continue to consider the possible risks and undesirable side-effects associated to cataract surgery, such as post-cataract endophthalmitis (POE), postcataract opacification (PCO), PCME, dysphotopsias, retinal detachment, and IOL dislocation.

DETAILED DESCRIPTION:
This is an observational, non-controlled, prospective clinical investigation to evaluate long-term safety and performance of Mini 4 Ready Intraocular Lenses in cataract patients.

Specifically the aim of the investigation is to evaluate:

* Accumulated incidence of surgical reinterventions and of achievement of visual acuity (VA) of 0.3 logMAR units or better after 1 and 2 years following IOL implant;
* Evaluation of contrast sensitivity (CS) after 1 month following IOL implant.
* Incidence and severity of posterior capsule opacification (PCO) and incidence of posterior capsulotomy after 1 and 2 years following IOL eye implant.
* Monocular and binocular uncorrected (UDVA) and corrected (CDVA)distance VA at 4 m under photopic conditions at 1 and 6 months.
* Overall refractive power, measured as manifest (subjective) and subjective refraction, standard and converted to spherical equivalent refraction at 1 and 6 months and at 1 and 2 years.
* Defocus curve of the implanted eye under photopic conditions at 1 month.
* Occurrence of surgical reinterventions for whichever reason.
* Occurrence of any adverse untoward outcome, including any adverse event (such as, but not limited to, pseudophakic cystoid macular edema (PCME), retinal detachment, signs of inflammation, surgical site infections (SSI), pupillary block, and IOL tilt and decentration).
* Accumulated incidence of surgical reinterventions and of achievement of visual acuity (VA) of 0.3 logMAR units or better after 1- and 6-months following index eye implant.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be deemed eligible for the study if all of the following inclusion criteria are met:

1. Older than eighteen years of age at the time of surgery and diagnosed with cataract;
2. Unilateral or bilateral cataract removal by phacoemulsification;
3. Correction of resulting aphakia with the Mini 4 Ready IOL. Indication for use of the Mini 4 Ready should be previous to and not conditioned by study participation.
4. In case of bilateral cataract, subject able to underwent second cataract surgery within 1 months from first implant and not before 7 days;
5. Willing and able to complete all required postoperative visits;
6. Able to comprehend and sign a statement of informed consent consistent with local regulation for research in human subjects.

Exclusion Criteria:

* Subjects participating in a concurrent clinical trial or who have participated in an ophthalmological clinical trial within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population comprise men and women aged ≥18 years requiring unilateral or bilateral cataract surgery and who are eligible for a monofocal IOL. The source population comprise patients scheduled to receive the Mini 4 Ready IOL in whom the cataractous lens could be removed by phacoemulsification following circular capsulorhexis, leaving the posterior capsule intact.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
surgical reinterventions and visual acuity (VA) 1-2 years | 1 - 2 years post implant
  Long-time accumulated incidence of surgical reinterventions and of achievement of visual acuity (VA) of 0.3 logMAR units or better after 1 and 2 years following IOL implant.

SECONDARY OUTCOMES:
contrast sensitivity | 1 month post implant
  Evaluation of contrast sensitivity (CS)
posterior capsule opacification (PCO) | 1 and 2 years post implant
  Incidence and severity of posterior capsule opacification (PCO)
posterior capsulotomy | 1 and 2 years post implant
  Incidence and severity of posterior capsulotomy
Monocular and binocular uncorrected (UDVA) | 1 and 6 months post implant
  Monocular and binocular uncorrected (UDVA) VA at 4 m under photopic conditions
Monocular and binocular corrected distance VA (CDVA) | 1 and 6 months post implant
  Monocular and binocular corrected distance VA (CDVA) at 4 m under photopic conditions
manifest refraction | 1 month, 6 months, 1 year and 2 years
  Overall refractive power, measured as manifest objective and subjective refraction, standard and converted to spherical equivalent refraction
defocus curve | 1 month
  Defocus curve of the implanted eye under photopic conditions
surgical reinterventions | 6 months
  Occurrence of surgical reinterventions for whichever reasons
adverse events | 6 months
  Occurrence of any adverse untoward outcome, including any adverse event (such as, but not limited to, pseudophakic cystoid macular edema (PCME), retinal detachment, signs of inflammation, surgical site infections (SSI), pupillary block, and IOL tilt and decentration).
surgical reinterventions and visual acuity (VA) 1 - 6 months | 1 and 6 months
  Short-time accumulated incidence of surgical reinterventions and of achievement of visual acuity (VA) of 0.3 logMAR units or better

CONTACTS AND LOCATIONS:
Locations (1):
- Daniela Nicolosi, Catania, Italy

IPD SHARING:
Plan to Share IPD: Undecided